CLINICAL TRIAL: NCT01668147
Title: Influence of Efavirenz and Ritonavir on Human Brain P-Glycoprotein Activity Using PET Imaging
Brief Title: Efavirenz and Ritonavir on Human Brain P-Glycoprotein
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 201205135
Record Dates: First submitted 2012-07-30; First posted 2012-08-17 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Drug Effects
Keywords: PET Imaging; Efavirenz; Ritonavir; [11C] desmethyl-loperamide; Healthy volunteers
MeSH Terms: interventions — N-demethylloperamide; Ritonavir; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Experimental): Session 1: Control (no pretreatment) - IV 10-14 mCi of [11C] desmethyl-loperamide (dLop) with PET/CT imaging
  Interventions: Drug: [11C] desmethyl-loperamide; Other: Control - no pretreatment
- Oral ritonavir (Active Comparator): Session 2: Pretreatment with oral ritonavir for 3 days followed by IV 10-14 mCi of [11C]dLop with PET/CT imaging
  Interventions: Drug: [11C] desmethyl-loperamide; Drug: Oral ritonavir
- Oral efavirenz (Active Comparator): Session 3: Pretreatment with oral efavirenz for 14 days followed by IV 10-14 mCi of [11C]dLop with PET/CT imaging
  Interventions: Drug: [11C] desmethyl-loperamide; Drug: Oral efavirenz

INTERVENTIONS:
Drug: [11C] desmethyl-loperamide — IV administration of 10-14 mCi of [11C] desmethyl-loperamide with PET/CT imaging
Other: Control - no pretreatment — Session 1: IV administration of 10-14 mCi [11C] desmethyl-loperamide (dLop) with PET/CT imaging and brain MRI
  Arms: Control
Drug: Oral ritonavir — Session 2: Pretreatment with oral ritonavir for 3 days followed by IV administration of 10-14 mCi [11C]dLop with PET/CT imaging and brain MRI
  Arms: Oral ritonavir
Drug: Oral efavirenz — Session 3: Pretreatment with oral efavirenz for 14 days followed by IV administration of 10-14 mCi [11C]dLop with PET/CT imaging and brain MRI
  Arms: Oral efavirenz

SUMMARY:
To determine the effects of ritonavir and efavirenz on the activity of P-glycoprotein in human brain.

DETAILED DESCRIPTION:
Sequential crossover using tracer 11C-desmethylloperamide, a substrate for brain P-glycoprotein, and positron emission tomography (PET), administered after nothing (control), oral ritonavir (3d), and oral efavirenz (14d) with washout in between

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female, 18-40 yr old
* Good general health with no remarkable medical conditions
* BMI < 33
* Provide informed consent

Exclusion Criteria:

* Known history of liver or kidney disease
* History of major medical conditions
* HIV seropositive
* Fasting blood glucose > 110 mg/dl
* Family history of type 2 diabetes
* Use of prescription or non prescription medications, herbals or foods known to be metabolized by or altering P-glycoprotein or CYP3A activity (hormonal birth control medications are acceptable if alternative means of contraception are used)
* Females who are pregnant or nursing
* Females taking hormonal contraceptives who are unwilling to use alternative means of contraception
* Contraindications to MRI
* Contraindications to PET scanning

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-08; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Kharasch, MD, PhD., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PET/CT Imaging: Session 1: Control (no pretreatment) - IV 10-14 mCi of [11C] desmethyl-loperamide (dLop) with PET/CT imaging Session 2: Pretreatment with oral ritonavir for 3 days followed by IV 10-14 mCi of [11C]dLop with PET/CT imaging Session 3: Pretreatment with oral efavirenz for 14 days followed by IV 10-14 mCi of [11C]dLop with PET/CT imaging
  [11C] desmethyl-loperamide: IV administration of 10-14 mCi of [11C] desmethyl-loperamide with PET/CT imaging after control, ritonavir or efavirenz
Period: Overall Study
Arm/Group | PET/CT Imaging
Started | 13
Completed | 7
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Groups:
- Study Arm: Session 1: Control (no pretreatment) - IV 10-14 mCi of [11C] desmethyl-loperamide (dLop) with PET/CT imaging Session 2: Pretreatment with oral ritonavir for 3 days followed by IV 10-14 mCi of [11C]dLop with PET/CT imaging Session 3: Pretreatment with oral efavirenz for 14 days followed by IV 10-14 mCi of [11C]dLop with PET/CT imaging
  [11C] desmethyl-loperamide: IV administration of 10-14 mCi of [11C] desmethyl-loperamide with PET/CT imaging after control, ritonavir or efavirenz
Arm/Group | Study Arm
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Cerebral [11C]dLop Distribution Volume
Time Frame: 1 day
Population: 0 Participants Analyzed/Assigned. The PI has left the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Groups:
- Control (no Pretreatment): Session 1: Control (no pretreatment) - IV 10-14 mCi of [11C] desmethyl-loperamide (dLop) with PET/CT imaging
  [11C] desmethyl-loperamide: IV administration of 10-14 mCi of [11C] desmethyl-loperamide with PET/CT imaging after control, ritonavir or efavirenz
- Oral Ritonavir: Session 2: Pretreatment with oral ritonavir for 3 days followed by IV 10-14 mCi of [11C]dLop with PET/CT imaging
  [11C] desmethyl-loperamide: IV administration of 10-14 mCi of [11C] desmethyl-loperamide with PET/CT imaging after control, ritonavir or efavirenz
- Oral Efavirenz: Session 3: Pretreatment with oral efavirenz for 14 days followed by IV 10-14 mCi of [11C]dLop with PET/CT imaging
  [11C] desmethyl-loperamide: IV administration of 10-14 mCi of [11C] desmethyl-loperamide with PET/CT imaging after control, ritonavir or efavirenz
Arm/Group | Control (no Pretreatment) | Oral Ritonavir | Oral Efavirenz
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Oral Ritonvir: Session 2: Pretreatment with oral ritonavir for 3 days followed by IV 10-14 mCi of [11C]dLop with PET/CT imaging
  [11C] desmethyl-loperamide: IV administration of 10-14 mCi of [11C] desmethyl-loperamide with PET/CT imaging after control, ritonavir or efavirenz
Arm/Group | Control (no Pretreatment) | Oral Ritonvir | Oral Efavirenz
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 2/13 | 4/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (no Pretreatment) (N=13) | Oral Ritonvir (N=13) | Oral Efavirenz (N=13)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Anxiety (Social circumstances) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes